CLINICAL TRIAL: NCT00051142
Title: A Safety and Efficacy Study of Travoprost 0.004% Compared to Latanoprost 0.005% in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: A Safety and Efficacy Study of Travoprost 0.004% Compared to Latanoprost 0.005% in Patients With Open-Angle Glaucoma (OAG) or Ocular Hypertension (OHT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-01-36
Record Dates: First submitted 2003-01-03; First posted 2003-01-07 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
Keywords: Glaucoma; POAG; OAG; OHT
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Travoprost; Latanoprost

INTERVENTIONS:
Drug: Travoprost
Drug: Latanoprost

SUMMARY:
The purpose of this study is to evaluate the safety and IOP-lowering efficacy of Travoprost (0.004%) compared to Latanoprost (0.005%) in patients with chronic open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Adult patients of any race and either sex with open-angle glaucoma (with or without pigment dispersion or pseudoexfoliation component) or ocular hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-02; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Investigators, Principal Investigator — Alcon Research
Locations (1):
- Latin America, Fort Worth, Texas, United States